CLINICAL TRIAL: NCT00213174
Title: School Playground Surfacing - A Randomized Prospective Comparison of Injury Rates on Sand Versus Wood Chip Surfaces
Brief Title: Study of Sand Versus Wood Chip Surfaces on School Playgrounds to Minimize Injury in School Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Andrew Howard, Interim Chief, Orthopaedics, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1000003531; CIHR: MCT-70318
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Wounds and Injuries; Closed Head Injury
Keywords: pediatrics; injury; arm fractures; trauma; playground surfaces; fractures
MeSH Terms: conditions — Wounds and Injuries; Head Injuries, Closed; Fractures, Bone

INTERVENTIONS:
Behavioral: school playgrounds

SUMMARY:
This study will compare children's injury rates (arm fracture, head injury and other injuries) when playing on playground equipment on granite sand versus wood fibre playing surfaces.

The hypothesis is that injury rates (arm fracture, head injury and other injuries) among school children are equal on granite sand and wood fibre playground surfaces.

ELIGIBILITY:
Inclusion Criteria:

* School children
* Ages 5-11
* Injured on falls from play equipment during supervised school hours

Exclusion Criteria:

* Children injured outside of supervised school hours

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2005-01

PRIMARY OUTCOMES:
Upper extremity fracture rates

SECONDARY OUTCOMES:
Fracture rates, upper extremity
Head injury rates
All injury rates

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Howard, MD, MSc, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada